CLINICAL TRIAL: NCT07112690
Title: Ganglion Impar Neurolysis for Radiation-Induced Pain During Anal Cancer Treatment
Brief Title: Ganglion Impar Neurolysis for the Improvement of Radiation-Induced Pain During Localized Anal or Perianal Skin Cancer Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jolinta Lin, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00008783; NCI-2025-03026 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00008783 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP6445-24 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Localized Anal Carcinoma; Localized Anal Margin Carcinoma; Stage 0 Anal Cancer AJCC v8; Stage I Anal Cancer AJCC v8; Stage II Anal Cancer AJCC v8; Stage IIIB Anal Cancer AJCC v8
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (ganglion impar neurolysis) (Experimental): Patients undergo ganglion impar neurolysis with fluoroscopy during week 4 of CRT on study.
  Interventions: Other: Electronic Health Record Review; Procedure: Fluoroscopy; Procedure: Ganglion Impar Neurolysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Procedure: Fluoroscopy — Undergo fluoroscopy
  Other Names: Radio Fluoroscopy; Radiographic Fluoroscopy; RF
Procedure: Ganglion Impar Neurolysis — Undergo ganglion impar neurolysis
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well ganglion impar neurolysis works to improve radiation-induced pain during the treatment of anal or perianal skin cancer that has not spread to other parts of the body (localized). Treatment for anal or perianal skin cancer includes giving chemotherapy and radiation therapy (CRT) at the same time. CRT is frequently associated with several side effects, including radiation-induced pain. Despite advances in radiation therapy delivery, patients may still experience side effects which can lead to treatment breaks or treatment discontinuation. Ganglion impar neurolysis is a type of nerve block procedure in which medicine is injected directly into or around a nerve to block pain. The location of the procedure is near the tail bone and the medicine numbs the nerves that are in charge of sensation in the skin by the buttocks and genitalia. This may improve radiation-induced pain in patients receiving CRT for localized anal or perianal skin cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the feasibility of ganglion impar neurolysis on decreasing pain in patients undergoing definitive CRT for anal cancer defined as decreasing unscheduled treatment breaks to a median of ≤ 3 days.

SECONDARY OBJECTIVE:

I. To track toxicities and patient-reported outcomes (PRO) during treatment including intervention of ganglion impar neurolysis.

OUTLINE:

Patients undergo ganglion impar neurolysis with fluoroscopy during week 4 of CRT on study.

After completion of study intervention, patients are followed up during the last week of radiation therapy and at 3-6 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have diagnosis of localized anal cancer or perianal skin cancer and have either initiated or about to initiated definitive chemotherapy and radiation therapy for their cancer

  * Patients who are consistently reporting pain scores of 5 or higher or reporting high pain interference or distress will be approached to participate in the study
* Age > 18 years. Given the rarity of anal cancer in children, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky > 60%)
* Life expectancy of greater than > 12 months
* Ability to understand and the willingness to sign a written informed consent document
* Inclusion of women and minorities: Both men and women and members of all races and ethnic groups are eligible for this trial
* Willingness and ability of the subject to complete the questionnaire
* Previous cancer diagnosis (such as colon or previously resected anal cancer) is permitted
* A diagnosis of HIV or immunocompromised status is permitted

Exclusion Criteria:

* Absolute neutrophil count less than 1500
* Platelet count less 80,000

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment breaks | Up to 6 weeks
Change in pain scores | At weeks 4, 6, and 18
  Will be assessed using pre- and pos-procedure pain scores as well as Patient Reported Outcomes Measurement Information System (PROMIS)-29 Profile version (v) 2.0 scale, PROMIS Neuropathic Pain Quality 5a questionnaire, and Pain Catastrophizing Scale.

SECONDARY OUTCOMES:
Patient reported outcomes | At weeks 4, 6, and 18
  Will be assessed using European Organization for Research and Treatment of Cancer Colorectal Cancer Specific Quality of Life Questionnaire and Anal Cancer Questionnaire.
Narcotic use | Up to 6 weeks
  Will be assessed using daily narcotic pain medication pill log.
Incidence of adverse events | Up to 18 weeks
  Will be assessed using Common Terminology Criteria for Adverse Events v5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jolinta Y. Lin, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Grady Health System, Atlanta, Georgia